CLINICAL TRIAL: NCT05672355
Title: Randomized Observer-Blinded Phase 2 Trial of COVID-19 Booster With GEO-CM04S1 or mRNA Vaccine in Patients With Chronic Lymphocytic Leukemia
Brief Title: A Vaccine Booster (GEO-CM04S1) for the Prevention of COVID-19 in Patients With Chronic Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 22416; NCI-2022-10303 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22416 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Chronic Lymphocytic Leukemia; COVID-19 Infection
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; COVID-19 | interventions — Specimen Handling; CVnCoV COVID-19 vaccine; COH04S1 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This trial is observer-blinded because the physical appearance of GEO-CM04S1 and mRNA vaccine may vary. The investigators, treating clinicians, participants, and other study staff, including the nurses involved in soliciting or recording of AEs, will be blinded through the day 112 visit.
  The study statisticians, pharmacists, and nurses who administer the vaccine injections will be unblinded. To avoid inadvertent unblinding of the participants at the time of injection, the syringe will be obscured from view by the nurse during injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (GEO-CM04S1) (Experimental): Patients receive GEO-CM04S1 vaccine IM on days 0 and 84 on study. Patients undergo blood sample collections throughout the study and are monitored for 1 year.
  Interventions: Procedure: Biospecimen Collection; Biological: Synthetic MVA-based SARS-CoV-2 Vaccine COH04S1
- Arm II (mRNA Covid-19 Vaccine) (Active Comparator): Patients receive mRNA vaccine injection IM on days 0 and 84 on study. Patients undergo blood sample collections throughout the study and are monitored for 1 year.
  Interventions: Procedure: Biospecimen Collection; Biological: mRNA COVID-19 Vaccine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: mRNA COVID-19 Vaccine — Given IM
  Other Names: COVID-19 mRNA Vaccine; mRNA-based COVID-19 Vaccine; SARS-CoV-2 mRNA Vaccine
  Arms: Arm II (mRNA Covid-19 Vaccine)
Biological: Synthetic MVA-based SARS-CoV-2 Vaccine COH04S1 — Given IM
  Other Names: COH04S1; SARS-CoV-2 Vaccine COH04S1; sMVA-based SARS-CoV-2 Vaccine COH04S1
  Arms: Arm I (GEO-CM04S1)

SUMMARY:
This phase II trial compares the effect of the GEO-CM04S1 vaccine with the current standard of care vaccine in preventing COVID-19 infections in patients with chronic lymphocytic leukemia (CLL). The GEO-CM04S1 vaccine uses a modified vaccinia virus (MVA) backbone that may be more effective at boosting COVID-19 immunity in patients with poor immune responses. MVA strongly induces T cell expansion (infection fighting blood cells) even in the background of a suppressed immune system, which is the case in the targeted CLL patient population. Using the GEO-CM04S1 vaccine may be more effective at preventing COVID-19 infection in patients diagnosed with CLL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Estimate the T cell-based immune response rate on day 56 post-injection of synthetic MVA-based SARS-CoV-2 vaccine COH04S1 (GEO-CM04S1) vaccine boost administered at 2.5x10^8 plaque-forming unit (PFU) or standard of care (SOC) vaccine administered as standard of care.

SECONDARY OBJECTIVES:

I. Evaluate the safety of single-dose vaccine boost based on moderate and unacceptable toxicities up to day 28 post-injection for the GEO-CM04S1 and SOC vaccines.

II. Estimate the T cell-based immune response rate at day 112 post-injection of GEO-CM04S1 vaccine at 2.5x10^8 PFU vs SOC severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) messenger ribonucleic acid (mRNA) vaccine administered as COVID-19 vaccine boosters.

III. Select the more promising vaccine to study further as a booster in patients with CLL.

IV. Evaluate SARS-CoV-2 S and N-specific Th1 vs Th2 polarization. V. Estimate the magnitude and durability of T-cell-based immune responses over a 12-month period.

VI. Estimate the levels and durability of SARS-CoV-2-specific IgG in a 12-month period.

VII. Evaluate levels of antibodies neutralizing SARS-CoV-2 in original strain and in variants of concern (VOC) based on the Centers for Disease Control and Prevention (CDC) definition using Spike-pseudotyped lentivirus.

VIII. Evaluate the overall safety profile during follow-up (12 months). IX. Estimate the incidence and severity of COVID-19 infection during follow-up (12 months).

EXPLORATORY OBJECTIVES:

I. Determine the SARS-CoV-2 variant by sequencing virus from polymerase chain reaction (PCR)-confirmed infected participants.

II. Evaluate activated/cycling and memory phenotype markers in SARS-CoV-2 stimulated T cells.

III. Estimate SARS-CoV-2-specfic serum IgA levels measured by enzyme-linked immunoassay (ELISA).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive GEO-CM04S1 vaccine intramuscularly (IM) on days 0 and 84 on study.

ARM II. Patients receive mRNA vaccine injection IM on days 0 and 84 on study.

Patients undergo blood sample collections throughout the study and are monitored for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 1
* Histologically confirmed diagnosis of CLL according to World Health Organization (WHO) classification
* Prior COVID-19 Vaccination (2 or more Pfizer or Moderna) with last injection >= 3 months prior
* Fully recovered from the acute toxic effects (except alopecia) to =< Grade 1 to prior anti-cancer therapy
* White Blood Cells (WBC) >= 1,000/mm^3 (To be performed within 14 days prior to Day 1 of protocol therapy)
* Platelets >= 50,000/mm^3 (To be performed within 14 days prior to Day 1 of protocol therapy)
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease) (To be performed within 14 days prior to Day 1 of protocol therapy)
* Aspartate aminotransferase (AST) =< 2.5 x ULN (To be performed within 14 days prior to Day 1 of protocol therapy)
* Alanine transaminase (ALT) =< 2.5 x ULN (To be performed within 14 days prior to Day 1 of protocol therapy)
* Creatinine clearance <1.5 ULN (To be performed within 14 days prior to Day 1 of protocol therapy)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (To be performed within 14 days prior to Day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 weeks after the last vaccine injection

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Known current SARS CoV-2 infection
* Prior Evusheld or other anti-SARS CoV-2 prophylaxis < 2 weeks prior
* Prior hematopoietic cell transplantation (HCT) or chimeric antigen receptor (CAR) T cell therapy within the previous year
* Systemic corticosteroids required for chronic conditions at doses > 0.5mg/kg/day prednisone equivalent within 7 days of enrollment
* Intensive cytotoxic therapies, T-cell depleting therapies, within 30 days of enrollment; however, patients with stable disease on maintenance therapies are allowed (See ConMeds for lists of acceptable and contraindicated therapies)
* Participants who have had a live vaccine =< 30 days prior to administration of any dose of study vaccine or subjects who are =< 2 weeks within administration of inactivated vaccines (e.g., influenza vaccine). Flu shots are allowed > 2 weeks before a study vaccine injection and > 2 weeks post study vaccine injection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent (e.g., egg allergies)
* Active infection not controlled on appropriate therapy
* History of adverse event with a prior smallpox vaccination
* History of pericarditis or myocarditis
* Any MVA vaccine or poxvirus vaccine in the last 12 months
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
T cell response | Baseline to day 56
  Assessed by >= 3-fold increase in S-specific or N-specific IFN-gamma-secreting T cells over baseline at day 56 (Primary Immune Analysis [PIA]), using Enzyme-linked Immunosorbent Spot (ELISPOT) assay to quantify SARS CoV-2 reactive T cells.
  * Note: Missing immune response will not be imputed. Missing immune response will be categorized as no for intent-to-treat analysis but will be excluded in per-protocol analysis.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) moderate toxicity (MOD) | From each injection to Day 28 post injection
  Grade 2 AEs (based on Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) probably or definitely attributable to vaccine boost, lasting >= 7 days. The primary toxicity analysis will be summarized in terms of type, severity, time of onset, duration, probable association with GEO-CM04S1 vaccine and reversibility or outcome.
Incidence of AEs unacceptable toxicity (UT) | From each injection to Day 28 post injection
  Grade 3-5 AEs (based on CTCAE version 5.0) probably or definitely attributable to vaccine boost. The primary toxicity analysis will be summarized in terms of type, severity, time of onset, duration, probable association with GEO-CM04S1 vaccine and reversibility or outcome.
Incidence of myocarditis or pericarditis | Up to 42 days following final injection of study vaccine (GEO-CM04S1 or standard of care [SoC] mRNA-CoV-2 vaccine)
  Any grade probably or definitely attributable to vaccine boost.
Incidence of serious adverse events (SAEs) | From each injection to Day 365 post injection
  At least possibly related to vaccine booster injection, with the exception of hospitalization for grades 1 or 2 fever.
T cell response | Baseline to 28 days after the second booster injection
  As assessed by >= 3-fold increase in S-specific or N-specific IFN-gamma-secreting T cells, using ELISPOT assay to quantify SARS CoV-2 reactive T cells. Scatterplots of immune response markers across time points will be generated to visualize the temporal patterns.
T cell fold-increase | At all immune test time points (Baseline, and days 28, 56, 84, 112, 180 and 365)
  ELISPOT assay of SARS CoV-2 reactive T cell cytokines (IFN-gamma, IL-4).
SARS-CoV-2-S and -N specific IFNgamma (Th1) and IL-4 (Th2) cytokine levels following stimulation with overlapping peptide libraries specific for SARS-CoV-2 | Up to 2 years
  The immune response rate at day 112 and 90% CI will be calculated by arm. Continuous immune response markers will be summarized by means or geometric means and standard deviations if the assumption of normal distribution is not violated. Repeated immune response measurements at the multiple time points will be analyzed using generalized estimating equations (GEE) or mixed regression models. Scatterplots of immune response markers across time points will be generated to visualize the temporal patterns.
Level of antibodies neutralizing SARS-CoV-2 Spike pseudoviruses | At day 56 after the first booster injection (PIA), at 28 days after the second booster injection (day 112), and at days 180 and 365
  Based on ancestral Wuhan strain and SARS-CoV-2 variants of concern (VOC) or variants of high consequence (VHC) based on Centers for Disease Control and Prevention (CDC) definition.
Levels of S- or N-specific IgG titers | At day 56 after the first booster injection (PIA), 28 days after the second booster injection (day 112), and at days 180 and 365
  Using quantitative enxyme-linked immunoassay (ELISA) based on World Health Organization (WHO) international standard for SARS-CoV-2 antibodies.
Confirmed COVID-19 infection by PCR viral load | Baseline to 1 year
Severe COVID-19 infection by Food and Drug Administration (FDA) criteria | Baseline up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alexey V Danilov, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States